CLINICAL TRIAL: NCT00710073
Title: Sono-Electro-Magnetic Therapy for the Treatment of Chronic Pelvic Pain Syndrome: A Pilot Study
Brief Title: Sono-Electro-Magnetic Therapy for Refractory Chronic Pelvic Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Thomas M. Kessler, MD, Department of Urology, University of Bern, 3010 Bern
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KEK99_06
Record Dates: First submitted 2008-07-02; First posted 2008-07-03 (Estimated); Last update posted 2008-07-03 (Estimated); Status verified 2008-07

CONDITIONS: Chronic Pelvic Pain Syndrome
Keywords: Chronic pelvic pain syndrome; Neuromodulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): Combined sono-electro-magnetic therapy
  Interventions: Device: sono-electro-magnetic therapy (Sonodyn Medico Star)

INTERVENTIONS:
Device: sono-electro-magnetic therapy (Sonodyn Medico Star) — twice a day for 10 minutes during 6 or 12 weeks
  Other Names: Sonodyn Medico Star

SUMMARY:
Treatment of chronic pelvic pain syndrome (CPPS) is challenging for patients and physicians once conventional therapies fail.

We hypothesize that combined sono-electro-magnetic therapy can improve refractory CPPS in men.

ELIGIBILITY:
Inclusion Criteria:

* CPSS III
* symptomatic >3 months
* NIH-CPSI total score =/>15
* NIH-CPSI pain =/>8

Exclusion Criteria:

* post void residual >100mL
* urinary tract infection
* urethral stricture
* age <18 years

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2006-05; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
National Institutes of Health Chronic Prostatitis Symptom Index (NIH-CPSI) | before treatment, after 6 weeks of treatment, if effective also after 12 weeks of treatment

SECONDARY OUTCOMES:
Pain visual analogue scale | before treatment, after 6 weeks of treatment, if effective also after 12 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Thomas M Kessler, MD, Principal Investigator — Department of Urology, University of Bern, 3010 Switzerland
Locations (1):
- Department of Urology, Bern University Hospital, Bern, Switzerland